CLINICAL TRIAL: NCT05377073
Title: Effects of Hatha Yoga vs Stretching in People With Mild to Moderate Parkinson's Disease
Brief Title: Effects of Complementary Therapies in People With Mild to Moderate Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Izaro Esain, Dr, Lecturer, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Esain I. Parkinson
Record Dates: First submitted 2022-05-09; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease
Keywords: Yoga; Stretching; Parkinson disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial
Who Masked: Investigator
Masking Description: Participants were randomly assigned (in a 1:1 ratio) through sealed opaque envelopes to either to the yoga group or the stretching group by coin tossing sequence generation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hatha Yoga (Experimental): Participants performed 1 hour supervised Yoga sessions once a week for a total of eight weeks.
  Interventions: Other: Hatha Yoga
- Stretching (Experimental): Participants performed 1 hour supervised Stretching sessions once a week for a total of eight weeks.
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Hatha Yoga — Patients in the yoga group performed warm-up exercises for 10 minutes, standing, sitting and supine positions of Hatha yoga (30 minutes), and relaxation and breathing exercises (20 minutes). The program consisted of one weekly session for a total of eight weeks.
  Arms: Hatha Yoga
Other: Stretching — Patients in the stretching group performed warm-up activities (10 minutes), and analytic stretching exercises targeting the following muscles: sternocleidomastoid, splenius, trapeze, triceps, posterior shoulder capsule, paravertebralis, hamstrings, quadriceps, gastrocnemius, soleus and tibialis anterior (40 minutes). Two repetitions of 15 seconds of each stretch were performed, with a 15 seconds interval between repetitions. The sessions ended with diaphragmatic breathing exercises (10 minutes). The program consisted of one weekly session for a total of eight weeks.
  Arms: Stretching

SUMMARY:
The aim of this study was to compare the effects of Hatha Yoga versus Stretching on physical outcomes, quality of life, physical activity and motor examination in persons with Parkinson Disease.

The hypothesis of this study is that Hatha Yoga will improve more than Stretching on physical outcomes, quality of life, physical activity and on motor examinations in persons with parkinson Diseases

DETAILED DESCRIPTION:
Individuals diagnosed with Parkinson 's disease, signed up at the Parkinson's association in Asparbi (Bilbao, Basque Country), and meeting the inclusion criteria were included in the study. These individuals were randomly assigned (in a 1:1 ratio) through sealed opaque envelopes to either to Hatha Yoga group and Stretching group by coin tossing sequence generation

Both programs consisted of one weekly session for a total of eight weeks.

Hatha Yoga group performed warm-up exercises for 10 minutes, standing, sitting and supine positions of Hatha yoga (30 minutes), and relaxation and breathing exercises (20 minutes).

Stretching group performed warm-up activities (10 minutes), and analytic stretching exercises targeting the following muscles: sternocleidomastoid, splenius, trapeze, triceps, posterior shoulder capsule, paravertebralis, hamstrings, quadriceps, gastrocnemius, soleus and tibialis anterior (40 minutes). Two repetitions of 15 seconds of each stretch were performed, with 15 seconds interval between repetitions. The sessions ended with diaphragmatic breathing exercises (10 minutes).

Demographic information form was filled out by patients including information about: age, height (cm), weight (kg). Additionally, the following measures are going to be measured:

* Postural control is assessed with a stabilometric platform.
* Flexibility ( Back Scratch Test and Chair Sit and Reach Test)
* Time Up and Go test (TUG)
* 5 Times Sit to Stand Test
* Walking speed
* Unified Parkinson´s Diseases Rating Scale III (UPDRS-III)
* International Physical Activity Questionnaires (IPAQ)
* Parkinson´s Disease Questionnaires- 39 (PDQ-39)

SPSS version 22 program was used in the analysis of the data. Mann Whitney U test, Wilcoxon test, Student T test and two-way mixed Anova were used to analyse the results.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of Parkinson's disease
* Stages I to III on the Hoehn and Yahr scale
* Ability to stand upright unaided and walk with or without technical support

Exclusion Criteria:

* Participate in another directed physical exercise program during the Project.
* Moderate or severe cognitive decline.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in height | 8 weeks
  Height is going to be assessed by portable stadiometer (Aisemed T226) to determine change from baseline.
Change from baseline in weight | 8 weeks
  Weight is going to be assessed by digital scale (Seca Model 868) to determine change from baseline.
Change from baseline in Postural control | 8 weeks
  Postural control, static balance is assessed with an stabilometric platform to determine change from baseline.
Change from baseline in Back Scratch Test | 8 weeks
  Flexibility of the upper limb is going to be assessed by the test of the Senior Fitness Test Back Scratch Test, to determine change from baseline.
Change from baseline in Chair Sit and Reach Test | 8 weeks
  Flexibility of the lower limb is going to be assessed by the test of the Senior Fitness Test Chair Sit and Reach Test, to determine change from baseline.
Change from baseline in Time Up and Go test (TUG) | 8 week
  Dynamic balance and agility is going to be assessed by Time Up and Go test to determine change from baseline.
Change from baseline 5 Times Sit to Stand Test | 8 weeks
  Lower limb strength is going to be assessed by 5 Times Sit to Stand Test to determine change from baseline.
Change from baseline in Walking speed | 8 weeks
  Walking speed is going to be assessed by walking 12 m, and photocells will be placed at 1 m and 11 m, recording time of 10 m to determine change from baseline.
Change from baseline in motor examination | 8 weeks
  Motor examination is going to be assessed by Unified Parkinson´s Diseases Rating Scale III to determine change form baseline. A higher score means a worse motor state. Total score subscale is 68.
Change from baseline in Physical Activity | 8 weeks
  Physical activity is going to be assessed by International Physical Activity Questionnaires to determine change from baseline. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (Metabolic equivalent of task minutes a week). Metabolic equivalent of task minutes represent the amount of energy expended carrying out physical activity.
Change from baseline in quality of life score | 8 weeks
  Quality of life score is going to be assess by Parkinson´s Disease Questionnaires- 39 to determine change from baseline. It has eight dimensions that are coded on a scale of 0 (perfect health as assessed by the measure) to 100 (worse health as assessed by the measure).

CONTACTS AND LOCATIONS:
Locations (1):
- University of the basque Country, Leioa, Bizkaia, Spain